CLINICAL TRIAL: NCT04005430
Title: A Phase I Study of Sequestered Transscleral, Controlled-Release Dexamethasone Delivered From an Episcleral Reservoir for Treatment of Macular Edema Secondary to Diabetes and Other Causes
Brief Title: A Phase I Study of Episcleral Dexamethasone for Treatment of Macular Edema
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Targeted Therapy Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3TDEX01
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Refractory Diabetic Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 1 (Experimental): Phase I open label study
  Interventions: Drug: Episcleral Dexamethasone

INTERVENTIONS:
Drug: Episcleral Dexamethasone — Sequestered Transscleral, Controlled-Release Dexamethasone
  Other Names: Sustained Release Transscleral Dexamethasone

SUMMARY:
This phase I trial will assess primarily the safety and secondarily anti-inflammatory effect of Episcleral Dexamethasone in patients suffering from refractory diabetic macular edema.

DETAILED DESCRIPTION:
This phase I trial will assess primarily the safety and secondarily anti-inflammatory effect of Episcleral Dexamethasone in patients suffering from refractory diabetic macular edema. Numerous studies have documented the anti-inflammatory activity of Dexamethasone in macular edema associated with diabetes, branch retinal vein occlusion, and non-infectious posterior uveitis. The investigators hypothesize that Episcleral Dexamethasone is safe, tolerable and that its anti-inflammatory activity will reduce macular edema and improve vision in patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Type I or II diabetes;
* Age >= 18 years;
* Visual acuity letter score in study eye < 70 and ≥ 25 letters (approximate Snellen equivalent 20/32 to 20/320);
* Ophthalmoscopic evidence of center-involved DME, within the central subfield (CSF);
* OCT CSF thickness value (microns):

  * Zeiss Cirrus: ≥290 in women; ≥305 in men
  * Heidelberg Spectralis: ≥305 in women; ≥320 in men
* Previous treatment with laser, anti-VEGF therapy and/or intravitreal steroids;
* No previous history of glaucoma or steroid-induced intraocular pressure response in either eye.

Exclusion Criteria:

* History of chronic renal failure requiring dialysis or kidney transplant;
* Retinal or optic nerve neovascularization on clinical exam, fundus photographs, or fluorescein angiograms;
* Evidence of external ocular infection;
* History of open-angle glaucoma or intraocular pressure >= 25 mmHg;
* History of steroid-induced IOP elevation that required IOP-lowering treatment;
* History of prior herpetic ocular infection;
* History of intravitreal or periocular corticosteroids within 3 months prior to enrollment;
* History of macular laser photocoagulation within 4 months prior to enrollment;
* History of antiangiogenic therapy within 4 weeks prior to enrollment;
* History of panretinal photocoagulation (PRP) within 4 months prior to enrollment or anticipated need for PRP in the next 6 months following enrollment;
* Presence of vitreomacular traction, epiretinal membrane, tractional retinal detachment, vitreous hemorrhage and or any ocular condition that the investigator judges could interfere in the safety and efficacy assessments;
* No other major non-diabetic pathology, or anticipation of such in the next 6 months following enrollment that in the opinion of the investigator would substantially and adversely affect assessment of safety and toxicity during the study;
* Participation in another clinical trial of non-approved medical treatment within 3 months prior to enrollment;
* Degenerative myopia;
* Malignant intraocular disease;
* Inability to understand informed consent, cooperate with testing or return to follow up visits; Pregnant or lactating women; Co-existent ocular disorder of the cornea, lens or media that will interfere with assessment of safety or efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure of the study is safety assessment. | 12 Months
  The main outcome of the study is safety assessment.

SECONDARY OUTCOMES:
Secondary outcomes are assessment of visual acuity. | 12 Months
  Secondary outcomes are assessment of visual acuity.
Secondary outcome are assessment of anatomical changes in the macula as measured via optical coherence tomography (OCT). | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Leng, MD, Principal Investigator — Stanford Medicine
Locations (1):
- Stanford Medicine Ophthalmology, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No